CLINICAL TRIAL: NCT00551356
Title: Comparison of the Insulin Therapies: Insulin Lispro Low Mix (25%) and Insulin Glargine in Patients With Diabetes Mellitus Type 2
Brief Title: Lispro Mix 25 vs. Glargine in Type 2 Diabetics
Acronym: IOOL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7354; F3Z-ME-IOOL
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes; Diabetic; Insulin; Humalog; Lantus; Glargine; Lispro
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — insulin lispro, isophane insulin lispro drug combination (25:75); Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Insulin glargine given SC once-daily in conjunction with oral antidiabetic medications.
  Interventions: Drug: Glargine
- 1 (Active Comparator): Lispro mix 25 SC twice-daily in conjunction with oral antidiabetic medications.
  Interventions: Drug: Insulin lispro mix 25

INTERVENTIONS:
Drug: Insulin lispro mix 25 — Insulin lispro mix 25 given SC twice-daily in conjunction with oral antidiabetic medications.
  Other Names: Humalog Mix25
  Arms: 1
Drug: Glargine — Insulin glargine given SC once-daily in conjunction with oral antidiabetic medications.
  Other Names: Lantus
  Arms: 2

SUMMARY:
In patients with type 2 diabetes who have not been on insulin therapy before the study will achieve better glycemic control by the treatment regiment consisting of two times daily insulin lispro mix 25 than by the treatment regiment with consisting of one time daily injection of insulin glargine. Improved glycemic control will be compared by the fasting plasma glucose and blood glucose excursions 2 hours after breakfast.

DETAILED DESCRIPTION:
The objective of this study is to investigate which type of insulin regimen is the best way to achieve best glycemic control in early type 2 diabetes. Patients with diabetes mellitus type 2 with a duration of diabetes between 1 and 10 years without previous insulin therapy will be randomized on insulin lispro mix 25 or insulin glargine therapy. Glycemic control will be compared by the between treatment difference in fasting plasma glucose and 2h postprandial blood glucose excursions (preprandial -postprandial excursions) after breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Males or females who have type 2 diabetes between 1 and 10 years
* Have used diet and/or maximum doses of oral antidiabetic agents (combination) for the treatment of their diabetes
* Have not been on insulin treatment within 3 months before entry into the study
* Have a hemoglobin A1c in the range of 8.0 to 12.5% according to a local laboratory within 4 weeks prior to or at Visit 1
* Have a body mass index below 40 kg/m²

Exclusion Criteria:

* Receive chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy (excluding topical and inhaled preparations) or have received such therapy within 2 weeks immediately prior to Visit 1
* Have a known allergy to insulin
* Have serum creatinine greater than or equal to 1.5 mg/dl as determined by a local laboratory
* Have known proliferative retinopathy
* Have had more than one unexplained episode of severe hypoglycemia (defined as requiring assistance of another person due to disabling hypoglycemia) within 6 months prior to entering the study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2002-11; Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline to endpoint in 2h postprandial blood glucose excursion after breakfast | 16 weeks or end of study.

SECONDARY OUTCOMES:
Hemoglobin A1c measured at endpoint | 16 weeks or end of study.
Change of hemoglobin A1c from baseline to endpoint | 16 weeks or end of study.
Glycemic control as determined by self-monitored blood glucose concentrations | 16 weeks or end of study.
The incidence and rate of self-reported hypoglycemic episodes | 16 weeks or end of study.
Body mass index (BMI) | 16 weeks or end of study.
Body weight | 16 weeks or end of study.
Total Insulin Doses | 16 weeks or end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City, Mexico

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com